CLINICAL TRIAL: NCT03549169
Title: Decision Making for the Management for the Symptoms in Adults of Heart Failure: Randomized Clinical Trial
Brief Title: Decision Making for the Management the Symptoms in Adults of Heart Failure
Acronym: TOMAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UNColombia
Record Dates: First submitted 2018-03-24; First posted 2018-06-07 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Heart Failure
Keywords: Intervention; Heart Failure; Symptoms management; Selft-care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: The participants are assigned to two groups during the duration of the study. A group receives the standard attention and the intervention protocol and the other group only the standard attention.
Who Masked: Outcomes Assessor
Masking Description: A research assistant (nurse trained in the measurement instruments) applies the instruments that allow the evaluation of the outcomes of interest: self-care, quality of life regarding health and follow up of clinical events: emergency attention, hospitalization, death by HF.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TOMAS (Experimental): Intervention centered on taking decisions for management of symptoms in adults with Heart Failure. Includes 3 doses (self-care maintenance, symptom perception and symptom management) and 4 strategies are developed: knowledge of the situation, experience and abilities in decision taking and compatibility with personal values.
  Interventions: Behavioral: TOMAS
- Standard or regular attention (Other): Regular attention is centered on education for therapeutic adherence
  Interventions: Behavioral: Regular attention

INTERVENTIONS:
Behavioral: TOMAS — Intervention focused on decision making for the management of symptoms aimed at adults with heart failure.
  Arms: TOMAS
Behavioral: Regular attention — Regular attention focused on education for therapeutic adherence
  Arms: Standard or regular attention

SUMMARY:
Introduction. Heart failure (HF) is the most prevailing chronic illness in the world. In Colombia, high morbidity and mortality rates because of HF are registered, as well as a significant burden of symptoms, frequent hospitalizations, poor quality of life, significant consumption of health resources and early mortality. It is necessary to propose novel strategies that can change the current picture.

Objective: determine the efficacy of an intervention centered in decision taking for the handling of symptoms in adults with HF who live in the department of Cordoba, Colombia.

Hypothesis

Primary hypothesis: the intervention Decision taking for the handling of symptoms in adults with HF: 1) Increases self-care.

Secondary hypothesis: 1) reduces clinical events: emergency care and hospitalizations, 3) Improves quality of life related to health.

DETAILED DESCRIPTION:
Intervention: The theoretic approach of the Theory of the Specific Situation Self-care in HF was used for the design of the intervention.

Supplier/dosage/duration. The intervention was given by the researcher (nurse trained in the intervention protocol) in three doses, each contact lasts 60 minutes. Frequency: sessions are given once a week during a one-month period (duration). Nurse controls are implemented after the intervention after one month and three months. There is also telephonic accompaniment on application of the participant.

Delivery method/environment. Verbal: Individual face to face. Printed educational written material type brochure, outpatient clinic of a health institution.

Methodology

Participants: inclusion criteria: adults (over the age of 18 years), more than two months of having been diagnosed; functional New York Heart Association (NYHA) Class II - III, left ventricular ejection fraction reduced (<40%). Cognitive state conservation (Lobo cognitive mini exam - MEC-35). Absence or low co-morbidity (Charlson index). Exclusion criteria: acute HF, advanced HF

Sample: The study was designed to have a 90% output, (alpha = 0.05), an expected difference of 0.5 in the outcome score of the management and maintenance evaluation in both groups, a standard deviation of outcome scores of 1.0, a correlation average between the first and the second evaluation of 0.2 and a rate of wear of 20%. Therefore, the required final sample size was 124 (62 per group - theoretic sample).

Pilot study: 176 adults with HF were recruited. 114 entered the study. 62 were excluded (did not meet the inclusion criteria (n=39), did not want to participate (=14), other reasons (n=9)).

Randomization. Table of random numbers without repetition. The Participants randomly assigned to the control group CG (n=57) received the standard attention, including standard education given by attention providers, and the ones assigned to the intervention group IG (n=57) received the intervention protocol.

Information collection (research assistant). The study registers information in the following time points: beginning (base line), follow up after a month (outpatient appointment), follow up after 3 months (outpatient appointment). The study is classified as simple blind; the research assistant, who is in charge of applying the instrument measuring the effect of the intervention, will remain blinded during the whole study regarding the group assigned to each participant.

Risk control. Compliance with methodological recommendations used to guarantee reliability and validity of the research studies proving a clinic intervention for behavioral changes. A plan is being contemplated that includes goals and strategies to monitor and counter possible threats to internal and external validity.

Ethical aspects. Compliance with universal ethical principles for research on humans, according to international ethical guidelines - CIOMS, national regulations, informed consent and deontological Nursing responsibilities in Colombia.

Analysis framework Excel database - SPSS Program analysis

1. Descriptive analysis of the total sample and by groups (intervention and control): absolute and relative frequency distributions; median and standard deviation.
2. Data normality analysis: Kolmogorov-Smirnov test Statistical analysis for independent samples a) difference of proportions: X2, b) difference of means: t for student, c) difference of medians: U test of Mann - Whitney. In all cases a statistic significance will be assumed if the value p < 0.05.
3. Intrasubject and intergroup analysis: ANOVA with repeated measurements.
4. Hypothesis proof: W of Mauchly test. When the sphericity premise is fulfilled, test F will be used.
5. Analysis of possible confusion and/or interaction effect.

   1. Stratified analysis: X2 of Mantel-Haenszel (M-H),
   2. Logistic regression analysis. Stepwise method. Minimum change % considered as favorable (≥20=1, ≤19=0).
6. Analysis of the magnitude of the intervention's effect. Improvement of at least 20% of the score on the scale, with the analysis principle of the intention of trying. The absolute increase in benefit and the necessary number for treatment (NNT) will be calculated afterwards.

ELIGIBILITY:
Inclusion criteria

* Adults (over 18 years of age).
* More than two months of having been diagnosed.
* Conserves cognitive state.
* Absence or low co-morbidity.

Exclusion criteria

* Confirmed diagnose of acute HF.
* Confirmed diagnose of advanced HF.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Self-care of heart failure index | Change from baseline self-care for heart failure index at 3 months
  The Self-Care of Heart Failure Index is a measure of self-care defined as a naturalistic decision making process involving the choice of behaviors that maintain physiologic stability and the response to symptoms when they occur. A score of ≥70 can be used as the cut-point to judge self-care adequacy.
  We strongly discourage users from calculating a total, combined SCHFI score. Instead, the data will be far more useful if the scales (maintenance, management, confidence) are used individually. Each scale is standardized to a score of 100.
  Use the following formula to compute a standardized:
  Maintenance: (sum of Section A items - 10) * 3.333 Management: (sum of Section B items - 4) * 5 Confidence: (sum of Section C items - 6) * 5.56

SECONDARY OUTCOMES:
Results in health | Change from baseline results in health at 3 months
  Emergency admissions, hospitalization, death by heart failure
Quality of life related to health | Change from baselineQuality of life related to health punctuation at 3 months
  The Minnesota Living with Heart Failure Questionnaire is one of the most widely used health-related quality of life questionnaires for patients with heart failure (HF). It provides scores for two dimensions, physical and emotional, and a total score. Comprising 21 items rated on six-point Likert scales, representing different degrees of impact of HF on quality of life related to health, from 0 (none) to 5 (very much). It provides a total score (range 0-105, from best to worst HRQoL), as well as scores for two dimensions, physical (8 items, range 0-40) and emotional (5 items, range 0-25). The other eight items (of the totalof 21) are only considered for the calculation of the total score.
  The Minnesota Living with Heart Failure Questionnaire has been translated into and validated in Spanish - Colombia.

CONTACTS AND LOCATIONS:
Overall Officials: EUGENIA HERRERA GUERRA, NURSE, Principal Investigator — Universidad Nacional de Colombia
Locations (1):
- Eugenia Herrera Guerra, Montería, Departamento de Córdoba, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Publication of articles derived from the main study
Supporting Information: Study Protocol, CSR
Time Frame: They will be available when the main study ends
Access Criteria: They will be available when the main study ends It can be requested by email

REFERENCES:
- See also: Riegel, B., Lee, C. S., Dickson, V. V., & Carlson, B. (2009). An Update on the Self-Care of Heart Failure Index. The Journal of Cardiovascular Nursing, 24(6), 485-497 — http://doi.org/10.1097/JCN.0b013e3181b4baa0
- See also: Riegel, B., Dickson, V., & Faulkner., K. (2016). The Situation-Specific Theory of Heart Failure Self-Care: Revised and Updated. The Journal of Cardiovascular Nursing, 31(3), 226-235. doi: 10.1097/JCN.0000000000000244 — https://journals.lww.com/jcnjournal/Abstract/2016/05000/The_Situation_Specific_Theory_of_Heart_Failure.7.aspx